CLINICAL TRIAL: NCT00671086
Title: A Phase 3, Open-label, Fixed-dose Study to Determine the Safety of Long-term Administration of TAK-375 in Subjects With Chronic Insomnia
Brief Title: Efficacy of Ramelteon in Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-02-TL-375-022; U1111-1114-3372 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Chronic Insomnia; DIMS (Disorders of Initiating and Maintaining Sleep); Disorders of Initiating and Maintaining Sleep; Insomnia Disorder Sleep Initiation Dysfunction; Transient Insomnia; Drug Therapy; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic | interventions — ramelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 16 mg QD (Experimental)
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — Subjects 65 yrs of age and older will take Ramelteon 8 mg, tablets, orally, once nightly for up to one year.
  Other Names: Rozerem; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Ramelteon — Subjects between 18 and 64 years of age will take Ramelteon 16 mg, tablets, orally, once nightly for up to one year.
  Other Names: Rozerem; TAK-375
  Arms: Ramelteon 16 mg QD

SUMMARY:
The purpose of this study is to determine the long-term safety of Ramelteon, once daily (QD), in subjects with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep or complaints of non-restorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is selective melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

The purpose of this study is to obtain data in support the safety of long-term use of Ramelteon for insomnia, and to determine whether there are any adverse effects associated with extended use. Participation in this study is expected to be about. Participation in this study is anticipated to be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria

* Participant has participated in an allowed Ramelteon study and has completed all final visit procedures for the previous study within 21 days of the Treatment Initiation Visit for this study.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Investigator believes that participant requires long-term treatment for insomnia.
* Primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised for at least 3 months and a history of daytime complaint(s) associated with disturbed sleep.
* Subjective sleep latency greater than or equal to 45 minutes and a subjective total sleep time less than or equal to 6.5 hours per night for at least 3 nights during the week of the Baseline Lead-in Period.
* Habitual bedtime is between 8:30PM and 12:00AM.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria

* Known hypersensitivity to Ramelteon or related compounds, including melatonin.
* Participated in any other investigational study, and/or taken any investigational drug within 30 days or five half-lives prior to Day 1 of study medication, whichever is longer. The only exception to this is prior participation in an allowed Ramelteon study.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to Day 1 of study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to Day 1 of study medication.
* Ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse with the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes 4 or more alcoholic drinks per day.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to Day 1 of study medication.
* Uses tobacco products during nightly awakenings.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study, or
  * not be in the best interest of the subject to participate in the study.
* Morning serum cortisol at the Baseline visit of less than 7.0 micro-g per dl.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Respiratory stimulants (eg, theophylline)
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Over-the-counter and prescription diet aids
  * Central nervous system active drugs
  * Narcotic analgesics
  * Beta blockers
  * St. John's Wort
  * Kava-kava
  * Gingko biloba
  * Melatonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1213 (Actual)
Dates: Start 2003-02; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events. | Week 1, Months 1, 2, 3, 4, 6, 8, 10, and 12 or Final Visit.
Change from Baseline in Vital Signs. | Week 1, Months 1, 2, 3, 4, 6, 8, 10, and 12 or Final Visit
Change from Baseline in Hematology Laboratory Tests. | Week 1, Months 1, 2, 4, 6, 8, 10, and 12 or Final Visit.
Change from Baseline in Chemistry Laboratory Tests. | Week 1, Months 1, 2, 4, 6, 8, 10, and 12 or Final Visit.
Change from Baseline in Urinalysis Laboratory Tests. | Week 1, Months 1, 2, 4, 6, 8, 10, and 12 or Final Visit.
Electrocardiograms. | Month 6 and 12 or Final Visit.
Menstrual Diary Results. | Week 1, Months 1, 2, 4, 6, 8, 10, and 12 or Final Visit.
Physical Examinations. | Months 2, 4, 8, 10, and 12 or Final Visit.

SECONDARY OUTCOMES:
Change from Baseline in Subjective Total Sleep Time. | Week 1, Months 1, 2, 3, 4, 6, 8, 10, 12, and 12 or Final Visit.
Change from Baseline in Subjective Sleep Latency. | Week 1, Months 1, 2, 3, 4, 6, 8, 10, 12, and 12 or Final Visit.
Clinical Global Impression Scale. | Months 6 and 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (122):
- United States (122):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Burbank, California
  - Cerritos, California
  - Irvine, California
  - La Jolla, California
  - La Mesa, California
  - Lafayette, California
  - Murrieta, California
  - Newport Beach, California
  - Northridge, California
  - Redlands, California
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Pueblo, Colorado
  - Wheat Ridge, Colorado
  - Wilmington, Delaware
  - Brandon, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Edgewater, Florida
  - Fort Lauderdale, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Blairsville, Georgia
  - Macon, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Libertyville, Illinois
  - Skokie, Illinois
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - Shawnee Mission, Kansas
  - Florence, Kentucky
  - Louisville, Kentucky
  - Paducah, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Bryan Pogue, Maryland
  - Chevy Chase, Maryland
  - Frederick, Maryland
  - Prince Frederick, Maryland
  - Rockville, Maryland
  - Newton, Massachusetts
  - Ann Arbor, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Hattiesburg, Mississippi
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - Wentzville, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Clementon, New Jersey
  - Lawrenceville, New Jersey
  - Newark, New Jersey
  - Toma River, New Jersey
  - Brooklyn, New York
  - Kingston, New York
  - Lake Success, New York
  - Rochester, New York
  - White Plains, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dublin, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Duncansville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Lafayette Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Bristol, Tennessee
  - Cordova, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Oakland, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
  - Wauwatosa, Wisconsin

REFERENCES:
- [Result] Richardson GS, Zammit G, Wang-Weigand S, Zhang J. Safety and subjective sleep effects of ramelteon administration in adults and older adults with chronic primary insomnia: a 1-year, open-label study. J Clin Psychiatry. 2009 Apr;70(4):467-76. doi: 10.4088/jcp.07m03834. Epub 2009 Mar 10. PMID 19284927
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI